CLINICAL TRIAL: NCT04094467
Title: CLASSICAL ANTAGONIST PROTOCOL IN COMPARISON WITH AGONIST STOP PROTOCOL IN Polycystic Ovary Symdrome WOMEN UNDERGOING Intra-cytoplasmic Injection TRIAL: a Randomized Controlled Trial
Brief Title: Comparison Between Two Different Protocols in Polycystic Ovary Symdrome Women Undergoing Intra-cytoplasmic Injection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCOS-ICSI
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — cetrorelix; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): the antagonist protocol group" where they will do intra-cytoplasmic injection using classical antagonist protocol
  Interventions: Drug: Cetrorelix
- control group (Active Comparator): "agonist stop/antagonist protocol group" where they will receive mid luteal agonist in the preceding intra-cytoplasmic injection cycle before starting classical antagonist protocol
  Interventions: Drug: Cetrorelix; Drug: Leuprolide Acetate

INTERVENTIONS:
Drug: Cetrorelix — 0.25 mg subcutaneous injection daily for 6 days
Drug: Leuprolide Acetate — 0.1 mg subcutaneous injection daily for 12 days
  Arms: control group

SUMMARY:
Stein and Leventhal were the first to recognize an association between the presence of polycystic ovaries and signs of hirsutism and amenorrhea (eg,oligomenorrhea, obesity), After women diagnosed with Stein-Leventhal syndrome underwent successful wedge resection of the ovaries, their menstrual cycles became regular, and they were able to conceive. As a consequence, a primary ovarian defect was thought to be the main culprit, and the disorder came to be known as polycystic ovarian disease.

ELIGIBILITY:
Inclusion Criteria:

1. Women under 35 years with polycystic ovary syndrome criteria
2. Normal male semen parameters
3. Normal tubes either by hysterosalpingography &/or laparoscopy
4. Free from other endocrine abnormalities

Exclusion Criteria:

1. NON polycystic ovary syndrome Criteria
2. More than 35 years
3. Abnormal semen parameters
4. Pathological tube& pelvic factor
5. Other endocrine disorders

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2019-12-07 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
The difference in clinical pregnancy rate in both groups | 6 weeks
  ultrasound detection of fetal heart pulsations

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt